CLINICAL TRIAL: NCT07085832
Title: Assessment of Cardiopumonary Resuscitation (CPR) Competency Among Healthcare Providers at the End of Advanced Life Support Training Course in Egypt
Brief Title: Assessment of Cardiopumonary Resuscitation (CPR) Competency Post ALS Course
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, ICU, Associate professor, National Hepatology & Tropical Medicine Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NHTMRI-9
Record Dates: First submitted 2025-06-22; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Chestcompressionadequacy
Keywords: CPR, metrics
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Pre-course assessment:
  Baseline measurement of CPR skills for two minutes cycle using a validated simulator by specialized adult feedback manikins e.g. Prestan CPR Feedback Manikins (i.e. built-in indicators for compression rate and depth) Intervention: Participants complete an ALS course, including theoretical and practical components focused on scenario based simulations for CPR and chest compressions.
  Post-course assessment:
  Immediate assessment at the end of the second day for CPR competency of 2 minutes cycle using the same simulator and the same parameters assessed pre-course.The scoring method is designed so that each item in the checklist is awarded zero or one point, with zero indicating lack of skill and one is indicating proficiency in the relevant area. Thus, participants' skills levels are determined and categorized.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPR competency pre and post ALS Course (Other): assessment of participants prior to initiation of ALS course
  Interventions: Other: Education (ALS provider course) in Egypt

INTERVENTIONS:
Other: Education (ALS provider course) in Egypt — Participants complete an ALS course, including theoretical and practical components focused on scenario based simulations for CPR and chest compressions.

SUMMARY:
to assess chest compression competency in healthcare providers following ALS training to identify areas for improvement and ensure high-quality CPR delivery.

DETAILED DESCRIPTION:
Assessment of certain CPR metrics will be done by the following approach;

Pre-course assessment:

Baseline measurement of CPR skills for two minutes cycle using a validated simulator by specialized adult feedback manikins e.g. Prestan CPR Feedback Manikins (i.e. built-in indicators for compression rate and depth), the following metrics will be followed and recorded:

1. Chest Compression Metrics:

   A. Compression Depth: at least 2 inches (5 cm) for adults, with a maximum of 2.4 inches (6 cm)3.

   B. Compression Rate: 100 to 120 compressions per minute3. C. Release (Recoil): Full chest recoil is essential to allow for effective venous return3.

   D. Hands-off time (Pause): Measured during the simulation, less than 10 seconds3.

   E. Chest Compression Fraction (CCF): Calculated as the ratio of the time spent performing compressions to the total time spent on CPR (including compressions, ventilations, and any pauses). Target will be ≥80%4.

   F. Compression Quality: An overall assessment (percentage shown by the feedback device) of the effectiveness of compressions, which may include depth, rate, and continuity.
2. Ventilation Metrics:

A. Tidal Volume: Target will be 400-700 mL of air for visible chest rise (in adults)3.

B. Ventilation Rate: 1 breath every 6 seconds (10 breaths per minute during continuous chest compressions for adults)3.

Intervention:

Participants complete an ALS course, including theoretical and practical components focused on scenario based simulations for CPR and chest compressions.

Post-course assessment:

Immediate assessment at the end of the second day for CPR competency of 2 minutes cycle using the same simulator and the same parameters assessed pre-course.The scoring method is designed so that each item in the checklist is awarded zero or one point, with zero indicating lack of skill and one is indicating proficiency in the relevant area. Thus, participants' skills levels are determined and categorized.

ELIGIBILITY:
Inclusion Criteria:

* Providers who will complete an ALS training course (two day-course).

Exclusion Criteria:

* Providers who will not complete ALS training course, those with physical limitations preventing effective chest compressions. Providers who will take immediate life support course (one day course), candidates attend from other courses to attend missed session and candidates who arrive late and cannot join the pre-course assessment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to assess CPR competency between ALS providers at the end of the ALS course if they will achieve the standard cutoff values and score. | two day course
  CCF%
The primary outcome is to assess CPR competency between ALS providers at the end of the ALS course if they will achieve the standard cutoff values and score. | Two day course
  Chest compression depth %

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - NHTMRI, Cairo
  - NHTMRI, EgRC, Cairo

IPD SHARING:
Plan to Share IPD: Undecided
results after acceptance for publication